CLINICAL TRIAL: NCT01940185
Title: A Post-Approval Study of the LINX® Reflux Management System
Status: Completed | Type: Observational
Sponsor: Torax Medical Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 3545
Record Dates: First submitted 2013-09-06; First posted 2013-09-12 (Estimated); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Gastroesophageal Reflux Disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- LINX device: Patients implanted with the LINX® Reflux Management System.
  Interventions: Device: LINX device

INTERVENTIONS:
Device: LINX device

SUMMARY:
A Post-Approval Study of the LINX® Reflux Management System in a prospective, multicenter, single-arm study, with patients as their own control to monitor the safety and efficacy of the LINX implant procedure and device in a post-approval environment to supplement existing safety and efficacy data.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a candidate for treatment with the LINX Reflux Management System
* Patient has provided written informed consent for participation in the post-approval study.
* Patient has indicated a willingness to comply with study requirements and the follow-up schedule and assessments.
* Patient has been diagnosed with GERD as defined by abnormal pH testing.
* Patient continues to have chronic GERD symptoms despite maximum medical therapy for the treatment of reflux.

Exclusion Criteria:

* Patients with suspected or known allergies to titanium, stainless steel, nickel, or ferrous materials.
* Known circumstances that would make it unlikely for the patient to complete follow-up through 60 months.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Gastroesophageal Reflux Disease (GERD) as defined by abnormal pH testing, and who continue to have chronic GERD symptoms despite maximum medical therapy for the treatment of reflux
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2012-06-30 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Reduction of total GERD-HRQL score | 6 months, 12 months, and annually to 60 months
  Successful reduction of ≥ 50% in the total GERD-HRQL as compared to baseline.
Serious, device-related adverse events | 60 months
  Reporting all serious device-related adverse events and summarizing by the number of events, the number of study patients with event, and the percent of study patients implanted with event. No formal statistical hypothesis tests will be conducted.

SECONDARY OUTCOMES:
Related Adverse Events | 120 months
  Incidence rate of of device- and/or procedure-related adverse events
pH Measurements | The secondary measurements will be evaluated at yearly interval to 120 months (esophageal pH not conducted at 72, 84, 96 and 108 months)
  Reduction from baseline in Total % time esophageal pH<4
Reduction of Symptoms | The secondary measurements will be evaluated at yearly interval to 120 months
  Reduction from baseline on Foregut Symptom Questionnaire (frequency and severity of heartburn and regurgitation, extra-esophageal symptoms and side effect profile). No formal statistical hypothesis tests will be conducted. Any statistical analyses will be primarily descriptive.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (19):
  - Keck Medical Center of Univeristy of Southern California, Los Angeles, California
  - University of California San Diego, San Diego, California
  - Swedish Medical Center/SurgOne, Englewood, Colorado
  - Albany Surgical, Albany, Georgia
  - Esophageal Institute of Atlanta, PC., Atlanta, Georgia
  - Candler Hospital, Savannah, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Beth Israel, Boston, Massachusetts
  - Cuyuna Regional Medical Center, Crosby, Minnesota
  - VIP Surg PLLC, Las Vegas, Nevada
  - University Hospitals Cleveland Medical Center - Geauga, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Allegheny Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Virginia Hospital Center, Arlington, Virginia
  - Swedish Medical Center, Seattle, Washington
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Froedtert and Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Result] Louie BE, Smith CD, Smith CC, Bell RCW, Gillian GK, Mandel JS, Perry KA, Birkenhagen WK, Taiganides PA, Dunst CM, McCollister HM, Lipham JC, Khaitan LK, Tsuda ST, Jobe BA, Kothari SN, Gould JC. Objective Evidence of Reflux Control After Magnetic Sphincter Augmentation: One Year Results From a Post Approval Study. Ann Surg. 2019 Aug;270(2):302-308. doi: 10.1097/SLA.0000000000002789. PMID 29697454